CLINICAL TRIAL: NCT01187550
Title: A Phase IV Open-label Study of Predictive Markers in Growth Hormone Deficient Pre-pubertal Children Treated With Saizen®
Brief Title: Predictive Markers in Chinese Growth Hormone Deficiency (GHD) Children Treated With Saizen®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27709
Record Dates: First submitted 2010-08-22; First posted 2010-08-24 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Dwarfism, Pituitary
Keywords: Dwarfism, pituitary; Growth hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

INTERVENTIONS:
Drug: Recombinant human growth hormone (r-hGH) — Recombinant human growth hormone (r-hGH) administered at dose of 0.033 milligram/kilogram (mg/kg) body weight (0.1 International Unit [IU]/kg body weight) per day by subcutaneous injection.
  Other Names: Saizen

SUMMARY:
This is an open-label, prospective, multicentric, non-comparative, non-randomized Phase IV interventional study in which subjects pre-diagnosed with Growth Hormone Deficiency (GHD) were treated for 4 weeks with Saizen to compare the response between GHD children born appropriate for gestational age (AGA) and those born small for gestation age (SGA) after 4 weeks of Saizen therapy.

DETAILED DESCRIPTION:
The response to growth hormone (GH) treatment, short-term as well as long-term, displays considerable inter individual variability. This is particularly evident for the endpoint of paediatric GH administration, that is (i.e.) the growth response, which is pronounced in children who are affected by GHD. This is an open-label, multicentric study in which subjects pre-diagnosed with GHD were treated for 4 weeks with Saizen. Two hundred fourteen GHD evaluable pre-pubertal subjects were planned to be recruited in approximately 9 sites in China. Demographic data, medical history, tanner stage, physical examination, body weight, height, bone age measurement, body mass index, review of baseline medications and procedures and blood sampling were performed at baseline visit, end of treatment visit (week 4) and at 4 week follow-up visit.

OBJECTIVES

Primary objective:

* To compare the response between GHD children born AGA and those born SGA after 4 weeks of Saizen therapy

Secondary Objectives:

* To explore the contribution of selected genes to the phenotype of GHD children
* To explore the impact of gene polymorphisms on the levels of specific serum biomarkers in GHD children after 4 weeks of Saizen therapy
* To explore the relationships between changes in gene expression and changes in serum biomarkers after 4 weeks of Saizen therapy and the spectrum of gene polymorphisms in GHD children

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with documented pre-established diagnosis of GHD with a GH peak response of <10 microgram/liter (mcg/L) with 2 GH stimulation tests, without priming with estradiol
* Subjects with SGA defined as birth weight and/or length at least 2 standard deviations (SDs) below the mean for gestational age
* Subjects with prepubertal status according to Tanner
* Subjects with pre-established history of normal thyroid function or adequate substitution for at least 3 months
* Subjects with weight for stature within the population specific normal range (>5th and <95th percentiles) for gender
* Subjects with willingness and ability to comply with the protocol for the duration of the study
* Subjects whose parents or guardians written informed consent given before any study-related procedure that was not part of the subjects normal medical care, with the understanding that the subject or parent/guardian might withdraw consent at any time without prejudice to future medical care. If the child was old enough to read and write, a separate assent form was given

Exclusion Criteria:

* Subjects who acquired GHD due to central nervous system tumor, trauma, infection, infiltration (documented by imaging), and history of irradiation or cranial surgery
* Subjects with previous treatment with GH, growth hormone releasing hormone (GHRH), anabolic steroids or any treatment affecting growth
* Subjects who had previous treatment with corticosteroids, except in case of topical or inhaled corticosteroid administration for atopic disease. Corticosteroids for hormonal substitution were also allowed if the condition and the treatment regimen had been stable for at least 3 months
* Subjects with severe associated pathology affecting growth such as malnutrition, malabsorption, or bone dysplasia
* Subjects with chronic severe kidney disease
* Subjects with chronic severe liver disease
* Subjects with chronic infectious disease
* Subjects with acute or severe illness during the previous 6 months
* Subjects with significant concomitant illness that would interfere with participation or assessment in this study
* Subjects who had active malignancy (except non-melanomatous skin malignancies that had undergone surgical excision and/or biopsy, diagnosis and treatment to resolution)
* Subjects with history or active idiopathic intra-cranial hypertension (benign intracranial hypertension or pseudo-tumor cerebri)
* Subjects with diabetes mellitus type I & II
* Subjects with any autoimmune disease
* Subjects who had previous screening failure in this study
* Subjects who had used an investigational drug or participated in another clinical study within the last 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 214 participants enrolled in the study, 1 participant could not be categorized as appropriate for gestational age (AGA) or small for gestational age (SGA) since weight and height at birth was not available.
Groups:
- Appropriate for Gestational Age (AGA): Participants in AGA group received Saizen (recombinant human growth hormone, r-hGH) subcutaneously (sc) at the daily dose of 0.033 milligram/kilogram (mg/kg) body weight for 4 weeks.
- Small for Gestational Age (SGA): Participants in SGA group received Saizen (r-hGH) sc at the daily dose of 0.033 mg/kg body weight for 4 weeks.
Period: Overall Study
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Started | 183 | 30
Treated | 175 | 30
Completed | 169 | 29
Not Completed | 14 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Other | 3 | 0
Not completed — Randomized but not treated | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA) | Total
Number analyzed (Participants) | 175 | 30 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 213 participants, data for baseline measure (age) was available for only 205 participants who were treated.
  years | 10.52 (3.844) | 9.39 (4.349) | 10.35 (3.931)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 213 participants, data for baseline measure (gender) was available for only 205 participants who were treated.
  Participants
    Female | 46 | 6 | 52
    Male | 129 | 24 | 153

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Insulin Like Growth Factor-1 Standard Deviation Score (IGF-1 SDS) Levels at Week 4
Description: Insulin Like Growth Factor-1 Standard Deviation Score (IGF-1 SDS) was calculated as logarithm (log) 10 actual value of IGF-1 - log 10 (mean reference value of IGF-1) divided by log10 reference standard deviation of IGF-1.
Time Frame: Baseline and Week 4
Population: The intent-to-treat (ITT) population set included all the participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: nanogram/millilter (ng/mL)
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Number analyzed (Participants) | 175 | 30
nanogram/millilter (ng/mL)
  Baseline | -2.04 (2.341) | -2.22 (2.390)
  Change at Week 4 | 1.38 (1.358) | 0.85 (1.257)
Statistical Analysis 1: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); Test type: Superiority or Other; p = 0.194, Wilcoxon rank sum test

2. Secondary Outcome: Change From Baseline in Insulin Like Growth Factor Binding Protein-3 (IGFBP-3) Levels at Week 4
Time Frame: Baseline and Week 4
Population: ITT population set included all the participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: microgram/mL (mcg/mL)
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Number analyzed (Participants) | 175 | 30
microgram/mL (mcg/mL)
  Baseline | 3.16 (1.386) | 2.57 (1.525)
  Change at Week 4 | 0.58 (0.869) | 0.51 (0.805)
Statistical Analysis 1: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); Test type: Superiority or Other; p = 0.752, Wilcoxon rank sum test

3. Secondary Outcome: Change From Baseline in Fasting Glucose at Week 4
Time Frame: Baseline and Week 4
Population: ITT population set included all the participants who received at least 1 dose of study medication. Here 'N' (Number of participants analyzed) signified those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: millimole/liter (mmol/L)
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Number analyzed (Participants) | 173 | 30
millimole/liter (mmol/L)
  Baseline | 4.83 (0.471) | 4.46 (1.106)
  Change at Week 4 | 0.17 (0.578) | 0.22 (0.886)
Statistical Analysis 1: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); Test type: Superiority or Other; p = 0.710, Wilcoxon rank sum test

4. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 4
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: picomole/L (pmol/L)
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Number analyzed (Participants) | 172 | 26
picomole/L (pmol/L)
  Baseline | 36.17 (74.575) | 23.58 (14.892)
  Change at Week 4 | 10.08 (81.674) | 12.04 (32.389)
Statistical Analysis 1: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); Test type: Superiority or Other; p = 0.265, Wilcoxon rank sum test

5. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) Test at Week 4
Description: HOMA-IR is used to assess insulin resistance and calculated by an empirical mathematical formula based on fasting plasma glucose and fasting plasma insulin levels. HOMA-IR = fasting plasma insulin (picomole/liter [pmol/L]) * fasting plasma glucose (millimole/liter [mmol/L]) divided by 22.5.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L*mmol/L
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Number analyzed (Participants) | 171 | 26
pmol/L*mmol/L
  Baseline | 7.91 (15.662) | 5.06 (3.290)
  Change at Week 4 | 2.96 (18.458) | 2.48 (6.527)
Statistical Analysis 1: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); Test type: Superiority or Other; p = 0.308, Wilcoxon rank sum test

6. Secondary Outcome: Change From Baseline in Lipid Profile at Week 4
Description: Total cholesterol, high-density lipoprotein (HDL)-cholesterol, low-density lipoprotein (LDL)-cholesterol and triglycerides levels were evaluated.
Time Frame: Baseline and Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Number analyzed (Participants) | 174 | 30
mmol/L
  Baseline (Total Cholesterol) | 4.16 (0.752) | 4.22 (0.833)
  Baseline (HDL-Cholesterol) | 1.56 (0.452) | 1.59 (0.443)
  Baseline (LDL-Cholesterol) | 2.18 (0.672) | 2.19 (0.709)
  Baseline (Triglycerides) | 0.99 (0.527) | 1.02 (0.638)
  Change at Week 4 (Total Cholesterol) | -0.28 (0.601) | -0.03 (0.612)
  Change at Week 4 (HDL-Cholesterol) | -0.10 (0.317) | 0.02 (0.329)
  Change at Week 4 (LDL-Cholesterol) | -0.24 (0.546) | 0.02 (0.502)
  Change at Week 4 (Triglycerides) | 0.12 (0.551) | -0.09 (0.831)
Statistical Analysis 1: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); For total cholesterol: Wilcoxon rank sum test was used to calculate p-value; Test type: Superiority or Other; p = 0.078, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); For HDL-cholesterol: Wilcoxon rank sum test was used to calculate p-value; Test type: Superiority or Other; p = 0.033, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); For LDL-cholesterol: Wilcoxon rank sum test was used to calculate p-value; Test type: Superiority or Other; p = 0.041, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Appropriate for Gestational Age (AGA) vs Small for Gestational Age (SGA); For triglycerides: Wilcoxon rank sum test was used to calculate p-value; Test type: Superiority or Other; p = 0.091, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until 4 weeks post drug administration. AEs are classified as pre-treatment, treatment-emergent and post-treatment.
Description: Pre-Treatment:Medical conditions present at initial study visit that did not worsen in severity or frequency during study;Treatment-Emergent: If onset date of AE was on or after the first dose date of the study medication; Post-Treatment: If the onset date of AE was post 4 weeks after drug administration for participants who completed the study.
Arm/Group | Appropriate for Gestational Age (AGA) | Small for Gestational Age (SGA)
Serious Adverse Events (participants affected / at risk) | 1/175 | 0/30
Other Adverse Events (participants affected / at risk) | 27/175 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Appropriate for Gestational Age (AGA) (N=175) | Small for Gestational Age (SGA) (N=30)
Appendicitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Appropriate for Gestational Age (AGA) (N=175) | Small for Gestational Age (SGA) (N=30)
Conjunctivitis (Eye disorders) | 1 | 0
Eye Oedema (Eye disorders) | 1 | 0
Ocular Hypertension (Eye disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Hyperhidrosis (General disorders) | 0 | 1
Injection Site Dermatitis (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 1
Liver Function Test Abnormal (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Skin Infection (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other